CLINICAL TRIAL: NCT06453811
Title: The Effect of a Self-Efficacy Theory-Based Spouse Participation Childbirth Preparation Program on Fear of Childbirth, Self-Efficacy, Mode of Delivery and Birth Outcomes: A Randomized Controlled Trial
Brief Title: The Effect of Spouse Participation Childbirth Preparation Program on Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Fatma Nur Duman, Research Assistant, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LHU_FND1
Record Dates: First submitted 2024-06-01; First posted 2024-06-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Fear of Childbirth; Childbirth Self-Efficacy; Mode of Delivery; Childbirth Preparation Program
Keywords: Self-Efficacy; Childbirth Preparation; Fear of Childbirth; Mode of Delivery; Spousal Support; Nursing

STUDY DESIGN:
Intervention Model Description: After meeting the couples, their eligibility for inclusion in the study will be assessed. Subsequently, couples who meet the inclusion criteria will be asked to read the informed consent form and provide verbal and written consent. Pre-tests will be administered to eligible couples, who will then be assigned to either the experimental group (Self-Efficacy Theory-Based Spouse Participation Childbirth Preparation Program) or the control group according to the block randomization list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): According to the block randomisation method, the couples who are included in the experimental group by applying the pre-test will be included in the programme in groups of 3-4 couples by planning the day and time they can participate in the programme. At the end of the sessions, the training guide reflecting the training content will be given to the couples and they will be asked to read it at home and do their homework by using the relevant parts of the guide. At the same time, these couples will continue their routine pregnancy controls in the hospital. It is planned to complete the trainings once a week, twice in total and for two weeks. After the trainings are completed, it is planned to send at least three reminders by text message until the calculated delivery date. Brochures and text message content related to the training content will be used in the reminder.
  Interventions: Other: Self-efficacy Theory-based Childbirth Preparation Program
- Control Group (No Intervention): No additional intervention will be provided to couples in the control group, and they will receive the routine care provided at the hospital. This routine care includes standard antenatal follow-ups, during which pregnant women and their spouses receive information about pregnancy and childbirth only during physician examinations.

INTERVENTIONS:
Other: Self-efficacy Theory-based Childbirth Preparation Program — According to the block randomisation method, the couples who are included in the experimental group by applying the pre-test will be included in the programme in groups of 3-4 couples by planning the day and time they can participate in the programme. At the end of the sessions, the training guide reflecting the training content will be given to the couples and they will be asked to read it at home and do their homework by using the relevant parts of the guide. At the same time, these couples will continue their routine pregnancy controls in the hospital. It is planned to complete the trainings once a week, twice in total and for two weeks. After the trainings are completed, it is planned to send at least three reminders by text message until the calculated delivery date. Brochures and text message content related to the training content will be used in the reminder.
  Arms: Experimental Group

SUMMARY:
The research is designed as a pre-test, post-test, parallel-group, randomized controlled study to examine the effect of a spouse-participated childbirth preparation program based on self-efficacy theory on fear of childbirth, self-efficacy, mode of delivery and outcomes. Participants will be allocated to experimental and control groups through block randomization. Participants in the experimental group will be enrolled in a two-session spouse-participated childbirth preparation program based on self-efficacy theory once a week, in addition to receiving routine care at the hospital. Participants in the control group will not receive any intervention, only routine care provided at the hospital.

DETAILED DESCRIPTION:
Nulliparous pregnant women and their spouses who apply to the obstetrics and gynecology clinic and outpatient clinic of the hospital where the research will be conducted will be assessed for eligibility according to the inclusion criteria, and informed consent will be obtained. Subsequently, prospective fathers will be given a Personal Information Form and the Fathers' Fear of Childbirth Scale; prospective mothers will be given a Personal Information Form, the Wijma Delivery Expectancy/Experience Questionnaire Version A, the Childbirth Self-Efficacy Inventory Short Form, and the Perception of Spousal Support in Pregnancy Scale as pre-tests. Couples will be allocated to the experimental or control group according to a block randomization list. Couples assigned to the experimental group will be included in a three-week program, attending a self-efficacy theory-based childbirth preparation program in groups of 3-4 couples, scheduled according to their availability. At the end of the sessions, the training guide reflecting the content of the training will be given to the couples and they will be asked to read it at home and do their homework by using the relevant parts of the guide. At the same time, these couples will continue routine pregnancy controls in the hospital. Routine pregnancy check-ups at the hospital include standard antenatal follow-ups, and pregnant women and their partners receive information about the pregnancy and labour process only during the medical examination. It is planned to complete the trainings once a week, twice in total and for two weeks. After the trainings are completed, it is planned to send at least three reminders by text message until the calculated delivery date. Brochures and text message contents related to the training content will be used in the reminder. After completing the training, the Fathers' Fear of Childbirth Scale, the Childbirth Self-Efficacy Inventory Short Form, and the Perception of Spousal Support in Pregnancy Scale will be administered again. Following childbirth, the Wijma Delivery Expectancy/Experience Questionnaire Version B will be completed by the mothers, and the birth process information form will be filled out by the researcher. Couples in the control group will undergo the same pre-test and post-test assessments as the experimental group. However, no additional intervention will be provided to these couples, and they will receive the same routine care as the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Couples must be 18 years of age or older,
* Couples should be able to read and write Turkish,
* The pregnant woman has never given birth before,
* The pregnant woman is at 28-30 weeks of gestation,
* The pregnancy is viable and singular,
* The pregnant woman does not have an established indication for caesarean section,
* Routine controls during pregnancy are carried out in the hospital where the study is conducted.

Exclusion Criteria:

* Pregnancy achieved by assisted reproductive techniques,
* Participating in a birth preparation programme other than the routine pregnancy check-ups at the hospital,
* Failure to attend any of the sessions in the childbirth preparation programme,
* Failure to communicate in the postnatal period (no response to at least 3 telephone calls)
* Development of any indication for caesarean section during pregnancy,
* The birth takes place in a health institution different from the hospital where the research will be conducted.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The Childbirth Self-Efficacy Inventory Short Form | The pre-test will be administered before randomisation and the post-test will be administered 15 minutes after the training is completed (on the same day).
  Measures the level of self-efficacy of expectant mothers in childbirth. The lowest score that can be obtained from the overall scale is 32 and the highest score is 320. The highest score obtained from the overall scale means that women's self-efficacy levels in childbirth are high (Ersoy & Kukulu, 2011).
Birth Process Information Form | It will be applied two hours after the expectant mother gives birth.
  This form inquires about the mode of delivery and intervention at birth. One of the primary outcomes of the research is mode of delivery.

SECONDARY OUTCOMES:
The Fathers' Fear of Childbirth Scale | The pre-test will be administered before randomisation and the post-test will be administered 15 minutes after the training is completed (on the same day).
  Measures the level of fear of childbirth in expectant fathers. The minimum score that can be obtained from the scale is 17 and the maximum score is 85. As the score increases, the level of fear of birth experienced by fathers also increases (Calpbinici vd., 2023).
The Wijma Delivery Expectancy/Experience Questionnaire Version A-B | The pre-test will be administered before randomisation and the post-test 2 hours after the delivery.
  Measures the level of fear of childbirth in expectant mothers. The minimum score that can be obtained from the scale is 0 and the maximum score is 165. As the score obtained from the scale increases, women's fear of childbirth also increases (Korukcu vd., 2012; Korukcu vd., 2016).
The Perception of Spousal Support in Pregnancy Scale | The pre-test will be administered before randomisation and the post-test will be administered 15 minutes after the training is completed (on the same day).
  Measures pregnant women's perceived partner support. A minimum of 16 and a maximum of 80 points can be obtained from the scale. A higher score means higher perceived spousal support (Yurdakul vd., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Gölbaşı, Ph.D., Study Director — Lokman Hekim University
Locations (1):
- Lokman Hekim University, Ankara, Söğütözü Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calpbinici P, Uzunkaya Oztoprak P, Terzioglu F, Ustun Y. The Fathers' Fear of Childbirth Scale: a Turkish validity and reliability study. J Reprod Infant Psychol. 2024 Jun;42(3):424-438. doi: 10.1080/02646838.2023.2225084. Epub 2023 Jun 13. PMID 37309993
- [Background] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Background] Korukcu O, Bulut O, Kukulu K. Psychometric Evaluation of the Wijma Delivery Expectancy/Experience Questionnaire Version B. Health Care Women Int. 2016;37(5):550-67. doi: 10.1080/07399332.2014.943838. Epub 2014 Oct 8. PMID 25119342
- [Background] Yurdakul M, Beşen MA, Alıcı, D. Development of the Perception of Spousal Support in Pregnancy Scale (PSSPS): Reliability and Validity Studies. Journal of Education and Research in Nursing. 2020; 17(1): 258-266.
- [Background] Ersoy Y, Kukulu K. Validity and Reliability Study of Self-Efficacy in Labour and Delivery Scale [Master's Thesis]. Akdeniz University. 2011.